CLINICAL TRIAL: NCT03068650
Title: Expanded Access (Compassionate Use) Treatment Protocol Rindopepimut (CDX-110)
Brief Title: Expanded Access (Compassionate Use) Treatment Protocol Rindopepimut
Acronym: CDX-110
Status: No longer available | Type: Expanded Access
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: CDX110-05
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-06

CONDITIONS: Recurrent GBM
MeSH Terms: conditions — Glioblastoma | interventions — rindopepimut

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: rindopepimut — Rindopepimut is an experimental cancer vaccine that may act to promote anti-cancer effects in patients who have glioblastoma multiforme (GBM) that expresses an EGFR mutation, called EGFRvIII. Data from, a randomized, controlled phase 2 study in patients with EGFRvIII positive progressive glioblastoma (the ReACT trial) suggested that vaccination with rindopepimut could improve survival. A randomized, controlled phase III study in patients with newly diagnosed EGFRvIII expressing GBM did not show a survival advantage from rindopepimut vaccination.

SUMMARY:
Celldex endeavors to make investigational products available to patients with life-threatening diseases who have exhausted other treatment options and where there is a reasonable expectation of benefit over risk. Requests for expanded access to rindopepimut in patients with EGFRvlll expressing recurrent glioblastoma will be considered.

ELIGIBILITY:
Inclusion Criteria:

* The patient has histologically confirmed relapsed or recurrent GBM.
* EGFRvIII expression in tumor tissue, as assessed by a central laboratory using the Celldex assay.
* Prior or planned therapy must include standard chemoradiation with temozolomide, unless the patient is not a candidate.
* Systemic corticosteroid therapy tapered to less than 4 mg of dexamethasone (or equivalent) per day.
* The patient does not have a known allergy or hypersensitivity to KLH, GM-CSF or yeast derived products, or a history of anaphylactic reactions to shellfish proteins.
* The patient does not have abnormal organ function, active autoimmune disease, active infections or additional concurrent conditions that would compromise the patient's ability to safely receive rindopepimut vaccine therapy.
* The patient is surgically sterile or post-menopausal, or, if of child-bearing potential, had a negative serum pregnancy test within the week prior to initiation of rindopepimut and is not nursing.
* Males and females of childbearing potential must agree to practice an effective form of contraception during the time from signing of informed consent through 28 days after the last dose of rindopepimut.
* The patient is able to read and understand, and has signed a patient informed consent form, which outlines the anticipated benefits and risks of treatment with rindopepimut.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult